CLINICAL TRIAL: NCT05186493
Title: Laparoscopic Robot-assisted Pelvic Exenteration for Pelvic Primary and Recurrent Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ebbe Billmann Thorgersen, Principal investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 286145
Record Dates: First submitted 2021-11-26; First posted 2022-01-11 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Locally Advanced Pelvic Cancer That Require Pelvic Exenteration
Keywords: robot-assisted; pelvic exenteration; minimally invasive surgery; locally advanced rectal and sigmoid cancers; localized central pelvic recurrence of cervical cancer or endometrial cancers; feasibility
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Locally advanced pelvic cancer that requires total pelvic exenteration (Experimental): Adult patients (>18 years) with locally advanced pelvic cancer that require pelvic exenteration considered eligible for robot- assisted minimally invasive surgery by the respective multidisciplinary teams
  Interventions: Procedure: robot-assisted total pelvic exenteration

INTERVENTIONS:
Procedure: robot-assisted total pelvic exenteration — Patients with locally advanced pelvic cancer that require pelvic exenteration considered eligble, are operated minimmally invasive robot-assisted

SUMMARY:
The Radium Hospital Oslo University Hospital Estimated date of first patient enrolled: 3rd quarter 2021 Anticipated recruitment period: 4 years Estimated date of last patient completed: 4th quarter 2025

Locally advanced pelvic cancer that requires total pelvic exenteration

Expected study-specific follow-up period per patient: 5 years according to standard follow-up for this patient group

Primary endpoint:

R0 resection rate (circumferential resection margin >1mm)

Secondary endpoints:

Rate of conversion to open surgery, peri- and postoperative complications, hospital length of stay, wound healing at 3 months follow-up, Quality of Life measured by EORTC Quality of Life Questionnaire C-30 preoperatively, at 3 months and 3 year follow-ups, disease-free survival, overall survival.

Diagnosis specific endpoints.

Open label observational study.

DETAILED DESCRIPTION:
Pelvic exenteration for locally advanced rectal cancer (LARC) and locally advanced sigmoid cancer LARC includes tumours threatening the mesorectal fascia or invading adjacent organs and structures (9). Locally advanced sigmoid cancer is defined as tumors extending through the colon wall with perforation and/or invasion of adjacent organs or structures (10). Surgical removal is the standard curative approach for these tumours, and achievement of complete tumour removal, or R0 resection, is prognostically important. The Residual tumour (R) classification defines R0 resection as having > 1 mm margin between the tumour and surrounding normal tissue, R1 resection as ≤ 1 mm margin, and R2 as local macroscopic residual tumour after resection (11). If R0 resection is achieved, the outcome for the patient is dramatically superior compared to when resection is incomplete. In a large study of 1291 LARC cases, the overall survival was 43 months in R0 cases compared to 21 months if R1 resection was achieved (12).

Neoadjuvant therapy including chemotherapy and (chemo) radiotherapy ((C) RT) has resulted in improved local control (13), presumably by increasing the rate of complete surgical tumour removal (14), when the patient is operated. Total radiation dose towards the pelvis are usually 25-50 Gy, often with concomitant fluoropyrimidine-based chemotherapy. Although the neoadjuvant radiotherapy improves prognosis (14), it also imposes challenges. The surgery itself might be difficult because of edema and fibrosis resulting in potentially involved margins, and the healing after surgery is impaired leading to increased postoperative morbidity. This holds true for all tumours in the pelvis that receive radiotherapy before surgery. Despite neoadjuvant therapy, tumours still often require resection of neighboring organs in order to achieve R0-resection.

First described in 1948, total pelvic exenteration can be defined as the removal of the bladder, removal of the prostate (in males), removal of the uterus or the vaginal vault and partial or total resection of the vagina (in females), and the removal of the rectum with or without the anus (15). Total pelvic exenteration is extensive surgery with reconstructions that include two stomas. Locally advanced rectal cancers and locally advanced sigmoid cancers with multiorgan involvement e.g. rectal cancer invading the prostate or the urinary bladder are candidates for total pelvic exenteration.

Pelvic exenteration for recurrent cervical and endometrial cancer previously treated with radiochemotherapy and selected cases of primary advanced vulva cancer For patients with gynecologic cancer, pelvic exenteration is sometimes the only available curative treatment. Particularly patients with recurrent cervical and endometrial cancer previously treated with chemoradiation are considered candidates for pelvic exenteration. Selected cases of primary advanced vulva cancer are also considered for more extensive pelvic surgery such as modified anterior or posterior pelvic exenteration. In Norway, pelvic exenteration for recurrent cervical cancer is centralized to the Department for Gynecologic Oncology at the Oslo University Hospital and annually, approximately 10-15 patients are treated with total pelvic exenteration. An ongoing project in our Institution evaluating the clinical outcome of 95 patients treated with open pelvic exenteration for one of the above mentioned diagnoses revealed that about 50 % of the patients developed at least one severe complication (grade 3 or above according to the contracted Accordion severity grading system of surgical complications). 87% had negative surgical margins on final histology, but after median follow up time of 3.2 years, 59% of the patients had relapsed. About a third of those were central/pelvic recurrences. The high complication rate warrants further improvement of the surgical technique and minimally invasive surgery has emerged as a promising approach for selected patients (16, 17). Recently, case reports utilizing laparoscopic robot-assisted surgery have been published (18, 19). The reports indicate satisfactory oncological results and less surgical morbidity compared to open surgery.

In many of the case reports on gynecological exenterations the reconstruction of the urinary tract is done extra-corporally. In our Institution, robot-assisted intra-corporal urinary diversion is well established. Thus, the robotic approach for pelvic exenterations is attractive and feasible in our multidisciplinary surgical group.

Study design Open label observational study. Study objectives This study is a feasibility study of laparoscopic robot-assisted total pelvic exenteration for pelvic cancers.

Feasibility will be assessed through:

1. Determining the R0 resection rate in included study patients
2. Assessment of conversion rate to open surgery
3. Assessment of perioperative and postoperative complications

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* locally advanced pelvic cancer that require pelvic exenteration
* eligible for robot- assisted minimally invasive surgery by the respective multidisciplinary teams, may be included in the study.

Exclusion Criteria:

* Any reason why the patient in the investigator's opinion is not suited for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of R0 resection | up to three months from surgery
  R0 resection in oncological surgery means resection with circumferential margin >1mm from the tumour. R0 resection is considered as an important predictor for outcome.

SECONDARY OUTCOMES:
Rate of conversion from laparoscopic robot-assisted to open surgery | peroperative
  a quality indicator and feasibility measure for the procedure
Rate and type of postoperative complications | 90 days
  Any complications within the first 90 days after surgery
Hospital length of stay | up to 4 weeks
  How long the patient stay in Hospital after surgery
Disease free survival | up to 5 years
  If the patient have any recurrent disease
Overall survival | up to 5 years
  If the patient is alive
Quality of Life measured with the validated EORTC Quality of Life Questionnaire C-30 measurement tool (QoL C-30) | Preoperative, and at 3, 6, 12 and 36 months
  Quality of Life measured before and on specific controles postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital The Radium Hospital, Oslo, Norway